CLINICAL TRIAL: NCT02974517
Title: The Application of Time-lapse System in IVF/ICSI: Can it be Beneficial to Final Pregnancy Outcome?
Brief Title: The Application of Time-lapse System in IVF/ICSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, 1st Affilated Hospital, Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU Time-lapse
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: the Application of Time-lapes System in IVF/ICSI
Keywords: time-lapes; IVF/ICSI; pregnancy outcome
MeSH Terms: interventions — Fetoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Time-lapse-Auto: All embryos are cultured in EmbryoScope®; embryo scores are evaluated on day 3 by KID Score system.
  Interventions: Device: EmbryoScope®
- Time-lapse-Manual: All embryos are cultured in EmbryoScope®; embryo scores are evaluated on day 3 by embryologist.
  Interventions: Device: EmbryoScope®
- Conventional Group: All embryos are cultured in our daily used incubators; embryo scores are evaluated on day 3 by embryologist.

INTERVENTIONS:
Device: EmbryoScope® — The intervention is EmbryoScope® versus conventional incubators.
  Groups: Time-lapse-Auto; Time-lapse-Manual

SUMMARY:
Nowadays, the rapid development of human assisted reproductive technology (ART) has provided many help for couples with fertility issues. Even take baby home rate has been increased dramatically in the past several decades; both clinicians and embryologists are still struggling to improve pregnancy rates. Among all the strategies that the embryologists have tried, much work has been done to find better embryo culture conditions and embryo quality evaluation system. Currently, most centers in the world, including ours, are still using conventional incubators and manual embryo scoring system. This traditional method has several limitations, such as unstable environment during culture, and embryo scores can be different judged by different embryologists. EmbryoScope® by Vitrolife is a newly developed time-lapse embryo culture and analysis system. It is user-friendly, and suited for routinely daily use. In addition, its KID Score system can help embryologist select high quality embryos quickly, which leads to an overall increase in pregnancy outcome in IVF/ICSI cycles. The aim of this prospective cohort study is to evaluate the use of EmbryoScope® in our center.

DETAILED DESCRIPTION:
All patients included into this study are divided into three groups:

1. Time-lapse-Auto: All embryos are cultured in EmbryoScope®; embryo scores are evaluated on day 3 by KID Score system.
2. Time-lapse-Manual: All embryos are cultured in EmbryoScope®; embryo scores are evaluated on day 3 by embryologist.
3. Conventional Group: All embryos are cultured in our daily used incubators; embryo scores are evaluated on day 3 by embryologist.

The aim is to compare IVF/ICSI outcomes, such as pregnancy outcome, fertilization rate, cleavage rate, high quality embryo rate, blastocyst formation rate, among these three groups.

ELIGIBILITY:
Inclusion Criteria:

* First IVF/ICSI cycle;
* With normal ovarian reserve(FSH < 10 mIU/mL; antral follicle count>5);
* Age under 38 years old;
* With normal uterine;
* Tubal factor infertility

Exclusion Criteria:

* Pre-implantation genetic diagnosis cycles;
* Oocyte donation or sperm donation cycles.

Ages: 22 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All embyros are from women undergoing IVF/ICSI in our center.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 5 weeks after embryo transfer
  5 weeks after embryo transfer, gestational sac with fetal heart present inside uterus

SECONDARY OUTCOMES:
2 pronucleus (2PN) fertilization rate | 48 hours after oocyte retrieved day
  Number of 2PN/Matured oocytes
Blastocyst formation rate | 6 days after oocyte retrieved day
  Number of Blastocysts/Number of day 3 embryos cultured to blastocyst
High quality embryo rate | 72 hours after oocyte retrieved day
  High quality embryos that deserve to be transferred or cryopreserved/ Clevaged embryos in total

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medical Center, 1st Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu YG, Lazzaroni-Tealdi E, Wang Q, Zhang L, Barad DH, Kushnir VA, Darmon SK, Albertini DF, Gleicher N. Different effectiveness of closed embryo culture system with time-lapse imaging (EmbryoScope(TM)) in comparison to standard manual embryology in good and poor prognosis patients: a prospectively randomized pilot study. Reprod Biol Endocrinol. 2016 Aug 24;14(1):49. doi: 10.1186/s12958-016-0181-x. PMID 27553622
- [Background] Lazzaroni-Tealdi E, Barad DH, Albertini DF, Yu Y, Kushnir VA, Russell H, Wu YG, Gleicher N. Oocyte Scoring Enhances Embryo-Scoring in Predicting Pregnancy Chances with IVF Where It Counts Most. PLoS One. 2015 Dec 2;10(12):e0143632. doi: 10.1371/journal.pone.0143632. eCollection 2015. PMID 26630267